CLINICAL TRIAL: NCT05215938
Title: Evaluation of Intra Organ Sodium Levels by Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-210-21
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-01

CONDITIONS: Image, Body; Sodium Disorder
Keywords: MRI; Sodium imaging; B1 field correction; Kidney circadian sodium level variation; Multi-organ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples to measure:
  Urinary albumin/creatinine excretion ratio, Na+, K+ and osmolarity. The laboratory analyses will be performed within seven days of collection and all urine samples will be eliminated afterwards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study I: Multi-organ sodium imaging with B1 field correction: The scan will be performed in four area of interests (AOFs) to acquire sodium level signal form the thigh, heart, kidneys, and brain. Between each AOF the sodium receive coil will be moved to cover the specific organ. Determination of the sodium imaging method robustness is performed with a series of MRI sequences.
  The scans at the four AOFs are repeated to evaluate repeatability. The scan time with repositioning of coils is approximately 15 min per station (total scan time 2 hours).
  If needed the participants are able to have a break between scan stations.
  Interventions: Diagnostic Test: MRI examination
- Study II: Circadian sodium level variation in the kidney measured with MRI: Participation requires one full day at the MR Centre. MRI scans will be performed three times at the same day within the following time periods: 6.30-8.00 am. (before breakfast), 12.30-14-00 pm. (after lunch) and 21.00-22.00 pm. (after dinner). The scan time is expected to be 30-40 min at each scan (three scans are performed on one examination day), which requires a total scan time ~1½ hours.
  Participants are not allowed to perform excessive physical exercise the day before and during the study day. Lighter physical exercise as walking, biking etc. is accepted. Alcohol consuming is not allowed the day before and during the study day. The participants can drink and eat as usual, but all fluid intake and urinations shall be documented in a liquid urination schedule. Blood pressure will be measured at each scan session and urine samples are collected just after each scan session to assess the osmolarity.
  Interventions: Diagnostic Test: MRI examination

INTERVENTIONS:
Diagnostic Test: MRI examination — The magnetic resonance imaging session will be performed in a clinical 3T MRI scanner (GE healthcare). A commercial human intent non-diagnostic RF coil (PulseTeq) will be used for 23Na MRI.
  The scanner, coils and sequences are regularly used in research projects and validated for the same safety requirements as routinely used in the clinic. Nevertheless, the complete MRI session will be performed in research mode to use the advanced options (limits the usage to non-diagnostic purposes).
  Participants will be placed in a supine position with coils covering the area of interest (AOF).
  MRI examination will be performed by trained personnel.

SUMMARY:
The investigators aim to implement an innovative imaging tool for detection of sodium level changes in-vivo with a clinical magnetic resonance (MR) scanner system. Conventionally, MR imaging (MRI) is performed with the use of proton imaging. Nevertheless, detection of other nuclei such as sodium (23Na) are possible with dedicated radio frequency sequences and radio frequency antennas tuned to the lower radio frequency of sodium. Non-invasive detection of sodium level changes has great potential as a precursor of organ deficiency and possible organ failure.

This project seeks to determine a robust method for detection and characterization of sodium levels with MRI. The sodium levels of the kidneys are known to change throughout the day. Therefore, an evaluation of the kidney circadian sodium level variation is performed.

In the proposed project, the investigators will scan two groups divided into two separate studies:

Healthy controls for optimization of imaging (n = 5, scanned twice) Healthy controls for comparison of circadian variation (n = 10, scanned triple on one day)

Sodium MRI could greatly improve the understanding and diagnostic capabilities of several medical conditions. If successful, the proposed project will serve as the groundwork for future clinical studies.

DETAILED DESCRIPTION:
Background

Magnetic resonance imaging is considered the gold standard medical imaging modality for soft tissue characterization. The basic approach of MRI is acquiring resonance signal of proton (1H) spins which is abundant in soft tissue. In general, MRI scanner radio frequency antennas (RF coils) only tuned to transmit and receive at the frequency of hydrogen for proton imaging; however, it is possible to transmit and receive on other frequencies to create resonance images of different molecules.

Acquisition of other nuclei is performed with MR spectroscopy (MRS) and spectroscopic imaging (MRSI). For in vivo applications, common MR-active nuclei are protons (1H), phosphorus (31P), carbon (13C), sodium (23Na), and xenon (129Xe). Protons are the most common due to their high gyromagnetic ratio and natural abundance in the human body. Sodium is the second most abundant of the magnetic resonance sensitive nuclei.

Sodium MRI allows non-invasive examinations of intra-organ sodium concentrations and handling in vivo. These are coupled to electrophysiological and metabolic processes crucial to life. The methods have been thoroughly investigated in laboratory settings but has never made the transition to the clinic due to the inherently low signal to noise of sodium MRI [1]. Imaging is often challenged by a gyromagnetic ratio of about 1/4th of proton making the signal-to-noise ratio (SNR) of 23Na MRI about 6000 times lower than that of proton MRI [2]. Nevertheless, recent years has seen a renewed interest in sodium MRI due to major technical advances of MRI scanner systems and receive coils [1].

In vivo measurements of sodium levels are of special interest for determination of the energy dependent Na+/K+-ATPase (the sodium-potassium pump) - an important physiological transport process of healthy cells [3]-[5]. A transport process which is affected in many clinical conditions involving tissue injury, edema, or necrosis resulting in an increase of total sodium level [6].

Recent studies of sodium levels in healthy subjects have shown circadian variation of several physiological processes e.g. urine output, blood pressure and kidney function [7], [8]. A decrease in sodium excretion at night is showed in humans [7] and renal handling of sodium level is reported to follow circadian variations in mice [9]. It is therefore important to evaluate sodium imaging robustness, possible bias due to circadian variation, and a possible effect of disruption in the circadian rhythms leading to development or progression of certain diseases.

This study aims to evaluate the circadian rhythm in healthy human kidneys. If a circadian change of sodium levels is proven, further investigations of sodium level in diseases such as kidney disease can be developed. The results from this study will provide valuable information for assessment of sodium levels in humans and will contribute to the diagnostic process of multiple disease.

Aim

Increased recognition of the circadian variation is needed as it may result in a foundation for improved understanding of disease processes in several clinical conditions.

The overall aim of this study is to implement and validate an imaging protocol for detection of sodium level changes in-vivo and determine circadian sodium level variations. This will be carried out in two separate studies:

Study I - Evaluation of sodium levels in thigh, heart, kidney, and brain:

The aim of the study is to evaluate sodium levels in thigh, heart, kidney, and brain with the use of magnetic resonance imaging in healthy human subjects.

This initial study will determine the robustness of the sodium specific imaging method in determination of human sodium levels in different MR challenging conditions and organs. The study will provide the needed information to create an optimal scanning protocol for sodium imaging.

Study II - Circadian variations of sodium levels in kidneys:

The aim of the study is to estimate circadian variations in the sodium gradient of the kidney with use of MRI in healthy volunteers, and to relate the MRI findings with the osmolarity proven in urine samples. The investigators hypothesize that the sodium level follows a circadian rhythm. If proven investigations of sodium level in kidney disease can develop. The investigators hypothesize that assessing the sodium level in humans will contribute to the diagnostic process of kidney disease in the future.

Materials and methods

MRI examinations:

The magnetic resonance imaging session will be performed in a clinical 3T MRI scanner (GE healthcare). A commercial human intent non-diagnostic RF coil (PulseTeq) will be used for 23Na MRI.

The scanner, coils and sequences are regularly used in research projects and validated for the same safety requirements as routinely used in the clinic. Nevertheless, the complete MRI session will be performed in research mode to use the advanced options (limits the usage to non-diagnostic purposes).

Participants will be placed in a supine position with coils covering the area of interest (AOF).

MRI examination will be performed by trained personnel.

Study I - MR protocol:

The scan will be performed in four AOFs to acquire sodium level signal from the thigh, heart, kidneys, and brain. Between each AOF the sodium receive coil will be moved to cover the specific organ. Determination of the sodium imaging method robustness is performed with the following MRI sequences. An initial localization scan followed by evaluation of the main magnetic field inhomogeneities (B0 field map). Hereafter the radio frequencies (RF) of the scanner is calibrated (amplitude and frequency) for optimal sodium imaging and an evaluation of the sodium coil is achieved (B1+ field map). Finally, the sodium specific sequence is applied. The B0 and B1 maps are applied in pre-processing to account for magnetic field imperfections and improve sodium imaging robustness.

The scans at the four AOFs are repeated to evaluate repeatability. The scan time with repositioning of coils is approximately 15 min per station (total scan time 2 hours).

If needed the participants are able to have a break between scan stations.

Study II - MR protocol:

The main outcome is 23Na MRI images of the sodium level in kidneys. Furthermore, the investigators will perform blood oxygen level dependent (BOLD) magnetic resonance imaging (MRI) to assess changes in renal oxygenation. The MRI examination also measures kidney size, T1, T2 relaxation assed by magnetic resonance fingerprinting (MRF), ADC (DWI), 23Na distribution (23Na MRI) and perfusion (pCASL).

The scan time is expected to be 30-40 min at each scan (three scans are performed on one examination day), which requires a total scan time ~1½ hours.

Study II - Examination day Participation requires one full day at the MR Centre. MRI scans will be performed three times at the same day within the following time periods: 6.30-8.00 am. (before breakfast), 12.30-14-00 pm. (after lunch) and 21.00-22.00 pm. (after dinner). Participants are not allowed to perform excessive physical exercise the day before and during the study day. Lighter physical exercise as walking, biking etc. is accepted. Alcohol consuming is not allowed the day before and during the study day. The participants can drink and eat as usual, but all fluid intake and urinations shall be documented in a liquid urination schedule. Blood pressure will be measured at each scan session and urine samples are collected just after each scan session to assess the osmolarity.

ELIGIBILITY:
Inclusion criteria:

Participants are eligible if they can provide informed consent and meet the following criteria:

* Healthy men and women aged 20-60 years.
* Five participants of each gender are required in study II, whereto, gender is not of importance in study I.
* Healthy is defined as no use of medicine besides from contraceptives and vitamins.

Exclusion criteria:

The participants are not eligible if they fulfill any of the following criteria:

* Exclusion criteria for the MRI are contraindication to MRI such as claustrophobia or the presence of a pacemaker or other implanted metallic device.
* Persons with circumference including arms > 160 cm. (MR scanner bore size)
* Pregnant women are not allowed to volunteer.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Healthy men and women in the ages of 20 to 60.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of intra organ sodium levels by magnetic resonance imaging | 6 months
  The overall aim of this study is to implement and validate an imaging protocol for detection of sodium level changes in-vivo and determine circadian sodium level variations. This will be carried out in two separate studies.

SECONDARY OUTCOMES:
Study I: Multi-organ sodium imaging with B1 field correction | 6 months
  The aim of the study is to evaluate sodium levels in thigh, heart, kidney, and brain with the use of magnetic resonance imaging in healthy human subjects.
  This initial study will determine the robustness of the sodium specific imaging method in determination of human sodium levels in different MR challenging conditions and organs. The study will provide the needed information to create an optimal scanning protocol for sodium imaging.
Study II: Circadian sodium level variation in the kidney measured with MRI | 6 months
  The aim of the study is to estimate circadian variations in the sodium gradient of the kidney with use of MRI in healthy volunteers, and to relate the MRI findings with the osmolarity proven in urine samples. We hypothesize that the sodium level follows a circadian rhythm. If proven by our study, investigations of sodium level in kidney disease can develop. We hypothesise that assessing the sodium level in humans will contribute to the diagnostic process of kidney disease in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- MR Research Centre, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
The study is performed on healthy subjects to evaluate sodium MR imaging feasibility. Even though results are of value to the field further studies would require inclusion of a patient group or an intervention.

REFERENCES:
- [Derived] Vaeggemose M, Schulte RF, Hansen ESS, Miller JJ, Rasmussen CW, Pilgrim-Morris JH, Stewart NJ, Collier GJ, Wild JM, Laustsen C. A Framework for Predicting X-Nuclei Transmitter Gain Using 1H Signal. Tomography. 2023 Aug 24;9(5):1603-1616. doi: 10.3390/tomography9050128. PMID 37736981
- [Derived] Rasmussen CW, Bogh N, Ringgaard S, Birn H, Vaeggemose M, Schulte RF, Laustsen C. Daytime Variation in Kidney Perfusion, Oxygenation, and Sodium Concentration Assessed by Multiparametric MRI in Healthy Volunteers. J Magn Reson Imaging. 2024 May;59(5):1603-1611. doi: 10.1002/jmri.28983. Epub 2023 Sep 1. PMID 37656067